CLINICAL TRIAL: NCT03841240
Title: The Central Venous Catheter Related Complications in Critically Ill Patients: A Prospective Study
Brief Title: The Central Venous Catheter Related Complications in Critically Ill Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2018ZZJHZX003
Record Dates: First submitted 2019-01-29; First posted 2019-02-15 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-01

CONDITIONS: Catheter Thrombosis; Catheter-Related Infections; Central Venous Catheter Related Bloodstream Infection; Central Venous Catheter Thrombosis
Keywords: catheter; thrombosis; infection; ultrasound; risk factor
MeSH Terms: conditions — Catheter-Related Infections; Upper Extremity Deep Vein Thrombosis; Thrombosis; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this prospective clinical study, the researchers investigate the incidence of catheter-related thrombosis and catheter-related infection during indwelling central venous catheterization in critically ill patients, and analyzed the risk factors for catheter-related complications and the relationship between catheter-related thrombi and catheter-related infections. The sample size is about 500.

DETAILED DESCRIPTION:
A prospective clinical trial is conducted. Five hundred participants who need to place central venous catheters admit to the Department of Critical Care Medicine of Zhujiang Hospital,Southern Medical University from February 2019. Ultrasound is used for screening catheter-related thrombosis, and catheter-related infections are diagnosed according to the Guidelines for the Diagnosis and Management of Intravascular Catheter-Related Infections. The primary outcome is the incidence of catheter-related thrombosis and catheter-related infections. The primary exposure factors are age, gender, APACHE II, RBC, Hct, PLT, FIB, D-dimer, PCT, blood glucose, anticoagulants, and vasoactive drugs, catheter type, tube placement, indwelling time, etc. Descriptive analysis is used for the incidence of various complications. T-test or non-parametric statistical test is used for single factor analysis of risk factors, chi-square test or Fisher's exact probability test is used for counting data. Multivariate analysis of risk factors and the relationship between complications are analyzed by logistic regression. Statistical analysis is performed with SPSS Statistics version 20.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old and <80 years old;
* Central venous catheter is required to be placed through the internal jugular vein, subclavian vein or femoral vein;
* Catheter placement is estimated to be ≥ 72 hours.

Exclusion Criteria:

* The central venous catheter has been placed before entering the department;
* There is obvious trauma or infection at the site of implantation;
* There is already a blood vessel thrombus in the site before implantation;
* Recently, deep vein thrombosis or catheter-related thrombosis has occurred.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comes from the five critical medical wards of Zhujiang Hospital , including integrated area, cardiovascular severe ward, respiratory severe ward, neurological severe ward and neurosurgical severe ward.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-02-19 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of catheter-related complications | Average 10 days
  The incidence of catheter-related thrombosis and infections

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Critical Care Medicine of Zhujiang Hospital,Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided